CLINICAL TRIAL: NCT01047904
Title: Performance and Reliability of the Acclarent Iontophoresis System for Anesthetizing the Tympanic Membrane in Healthy Volunteers
Brief Title: Anesthetizing the Tympanic Membrane in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Integra LifeSciences Corporation (Industry)
Collaborators: Acclarent (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPR005006
Record Dates: First submitted 2010-01-11; First posted 2010-01-13 (Estimated); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Evaluate Performance and Reliability of Iontophoresis System

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Iontophoresis-treated (Experimental): Healthy volunteers will evaluate reliability and performance of Iontophoresis System in delivery of local anesthesia to the TM.
  Interventions: Device: Acclarent Iontophoresis System

INTERVENTIONS:
Device: Acclarent Iontophoresis System — Administration of local anesthesia using the Acclarent Iontophoresis System

SUMMARY:
The study will evaluate the performance and reliability of minor design changes to the Acclarent Iontophoresis System components for anesthetizing the tympanic membrane in healthy volunteers. Data collected from this study will enable the development of future applications and technology.

ELIGIBILITY:
Inclusion Criteria:

1. >=18 years of age
2. Both male and female subjects are eligible.

Exclusion Criteria:

1. Pregnant or lactating females
2. Subjects with a history of sensitivity or reaction to lidocaine, epinephrine or any hypersensitivity to local anesthetics of the amide type, or any component of the drug solution.
3. Markedly atrophic TM
4. Perforated TM
5. Sclerotic TM
6. Otitis externa
7. Electrically sensitive subjects and subjects with electrically sensitive support systems (pacemakers, defibrillators, etc.)
8. Damaged or denuded skin in the auditory canal
9. Cerumen impaction resulting in a significant amount of cleaning required to visualize the tympanic membrane
10. Evidence of Otitis Media at day of procedure, or within the past three (3) months prior to procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-08; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Procedural Success | X days
  Evaluation of the performance and reliability of the Acclarent Iontophoresis System in delivery of local anesthesia to the TM in healthy volunteers

SECONDARY OUTCOMES:
Incidence of adverse effects associated with the System and the Iontophoresis procedure | X days
  The investigator will rate any adverse event that occurs during the procedure for level of severity and relationship to the study device.
Tolerability of the iontophoresis system | X days
  Subject tolerability of the iontophoresis procedure will be assessed using a pain scale

CONTACTS AND LOCATIONS:
Locations (1):
- East Palo Alto, California, United States